CLINICAL TRIAL: NCT03032393
Title: The Effects of Posture on Timed up and go
Brief Title: The Effect of Power Posing on Timed Up and Go Test Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Weiqing Ge, Associate Professor, Youngstown State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 071-2017
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dominant (Experimental): Subjects in the experimental group were instructed to stand with hands on their hips, elbows pointing out and feet approximately one foot apart for 20 seconds.
  Interventions: Other: high-power
- Submissive (Active Comparator): Subjects in the control group were instructed to stand with hands and arms wrapping around the torso and feet together for 20 seconds.
  Interventions: Other: low-power

INTERVENTIONS:
Other: high-power — Subjects will stand with hands on their hips, elbows pointing out and feet approximately one foot apart (high-power) for 20 seconds.
  Arms: Dominant
Other: low-power — Subjects will stand with hands and arms wrapping around the torso and feet together (low-power) for 20 seconds.
  Arms: Submissive

SUMMARY:
This study determines the effects of posture on time up and go test. Half of the subjects will assume a high-power posture, while the other half will assume a low-power posture.

DETAILED DESCRIPTION:
Subjects in the experimental group were instructed to stand with hands on their hips, elbows pointing out and feet approximately one foot apart for 20 seconds. Subjects in the control group were instructed to stand with hands and arms wrapping around the torso and feet together for 20 seconds. Timed Up and Go test was administered using an OmniVR™ Virtual Rehabilitation System before and after the postural intervention

ELIGIBILITY:
Inclusion Criteria:

* male or female, age 18 to 65, with all 4 extremities intact, and ability to stand still for 20 seconds.

Exclusion Criteria:

* unable to stand with their feet together or one foot apart for at least 20 seconds, unable to wrap their arms around their torso or keep their hands on their hips for 20 seconds, unable to perform sit to stand transfer and ambulation independently, and cognitive impairments that interfere with the experimental procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hripko, Study Director — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dominant | Submissive
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dominant | Submissive | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Timed up and go Test
Description: Patients wear their regular footwear and can use a walking aid if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters or 10 feet away on the floor. The timed up and go test measures the amount of time, in seconds, that it takes to stand from a chair, walk 3 meters, turn around and walk back to the chair, and sit down again.
  A change between pre and post postural intervention is reported. The time point for pre intervention is at baseline. The time point for post intervention is immediately after the intervention.
Time Frame: Up to 3 minutes during each Timed up and go Test. Twice (pre and post the postural intention) at the same session (day).
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Dominant | Submissive
Number analyzed (Participants) | 15 | 15
second | -0.17 (0.65) | 0.20 (0.43)

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected for 11 months and 3 days during period of the data collection. For each participant, adverse event will be assessed for 1 day when the data collection is taken.
Arm/Group | Dominant | Submissive
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Limitations of the study included convenience sampling and the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03032393/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03032393/Prot_SAP_001.pdf